CLINICAL TRIAL: NCT03500159
Title: A 12-Week, Randomized, Multi-Center, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 2 Trial to Evaluate the Efficacy and Safety of AQX-1125 (200 mg) in Male Subjects With Chronic Prostatitis/Chronic Pelvic Pain Syndrome
Brief Title: Efficacy and Safety of AQX-1125 in Subjects With Chronic Prostatitis/Chronic Pelvic Pain Syndrome
Acronym: CP/CPPS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's Decision
Sponsor: Aquinox Pharmaceuticals (Canada) Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AQX-1125-205
Record Dates: First submitted 2018-04-04; First posted 2018-04-17 (Actual); Results first posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Chronic Prostatitis; Chronic Pelvic Pain Syndrome
MeSH Terms: interventions — 4-(4-(aminomethyl)-7a-methyl-1-methylideneoctahydro-1H-inden-5-yl)-3-(hydroxymethyl)-4-methylcyclohexan-1-ol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AQX-1125 (Experimental): AQX-1125 200 mg
  Interventions: Drug: AQX-1125 200 mg
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AQX-1125 200 mg — Synthetic SHIP1 activator
  Other Names: Rosiptor
  Arms: AQX-1125
Drug: Placebo — Appearance and weight matched tablets without the active product ingredient
  Arms: Placebo

SUMMARY:
This is a randomized, multi-center, double-blind, parallel-group study, enrolling approximately 100 male subjects diagnosed with CP/CPPS to evaluate the effect of 12-week treatment with AQX-1125 (active drug) compared to placebo.

The subjects will be randomized to receive orally once-daily either AQX-1125 (200 mg) or placebo in a 1:1 ratio across approximately 30 centers in North America (United States and Canada). The study will consist of a screening period of up to 3 weeks, a 12-week treatment period followed by a 4-week off drug safety follow-up period, and an ophthalmic safety follow-up call at 3 months and visit at 6 months post last dose, for a total study duration of about 41 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent and the willingness and ability to comply with all aspects of the study requirements
* Males, ≥18 and ≤80 years of age at Screening Visit 1
* Have pain or discomfort in the pelvic region for at least 3 months in the last 6 months, in the absence of a urinary tract infection or other pelvic/urological cause, and have a physician diagnosis of CP/CPPS (NIH Prostatitis Category III)
* Subjects must agree to use a condom for sexual intercourse from Screening Visit 1 until at least 90 days after the last dose of study drug, unless they have been surgically sterilized (vasectomy) for a minimum of 6 months
* Must be capable of voiding independently for 30 days prior to screening

Exclusion Criteria:

* Diagnosis of NIH Prostatitis Categories I (acute prostatitis) or II (chronic bacterial) prostatitis
* Diagnosis of interstitial cystitis/bladder pain syndrome (IC/BPS) with symptoms of pain, pressure, or discomfort perceived to be related to the bladder, and associated lower urinary symptoms for >6 weeks in the absence of infection or other identifiable causes
* Relief of pelvic pain after voiding
* Post-void residual volume >150 mL
* Have had an unresolved (positive bacterial urine culture) urinary tract infection within 8 weeks (inclusive) prior to Screening Visit 1
* History of previous prostate or bladder intervention within 1 month of Screening Visit 1, history of microwave therapy, transurethral resection of the prostate, transurethral radiofrequency thermotherapy, transurethral incision of the prostate, transurethral needle ablation, transurethral laser vaporization of the prostate, Urolift®, Rezum, and other urological interventions within 6 months of Screening Visit 1
* Unilateral testicular or scrotal pain as the sole symptom of CP/CPPS
* Ongoing, symptomatic urethral stricture disease
* Neurologic disease or disorder affecting the bladder, ability to void spontaneously, or directly contributing to urinary symptoms (e.g., multiple sclerosis, autonomic neuropathy)
* Severe, excruciating pain during rectal exam (i.e. an "inability to perform the exam")
* History of chronic substance abuse, dependency or abuse of opiates, or other narcotics within the last 2 years
* Any prior history of pelvic cancer (e.g., colorectal, genitourinary) or treatment (radiation or chemotherapy) thereof
* Major surgery within 3 months prior to Screening Visit 1
* Have any other condition/disease which, in the opinion of the Investigator, could compromise subject safety or interfere with the subject's participation in the study or in the evaluation of the study results.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 3 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Shoskes, MD, Principal Investigator — The Cleveland Clinic
Locations (27):
- United States (23):
  - Site 1026, Homewood, Alabama
  - Site 1010, Mobile, Alabama
  - Site 1004, Tucson, Arizona
  - Site 1028, Laguna Hills, California
  - Site 1018, Los Alamitos, California
  - Site 1016, Los Angeles, California
  - Site 1020, Los Angeles, California
  - Site 1027, New Port Richey, Florida
  - Site 1013, Coeur d'Alene, Idaho
  - Site 1015, Springfield, Illinois
  - Site 1023, Jeffersonville, Indiana
  - Site 1014, West Des Moines, Iowa
  - Site 1012, Shreveport, Louisiana
  - Site 1002, Royal Oak, Michigan
  - Site 1011, Albuquerque, New Mexico
  - Site 1009, Lake Success, New York
  - Site 1021, Charlotte, North Carolina
  - Site 1008, Raleigh, North Carolina
  - Site 1019, Wilmington, North Carolina
  - Site 1001, Cleveland, Ohio
  - Site 1017, Oklahoma City, Oklahoma
  - Site 1007, Philadelphia, Pennsylvania
  - Site 1022, Dallas, Texas
- Canada (4):
  - Site 1005, Brampton, Ontario
  - Site 1025, Kingston, Ontario
  - Site 1003, Oakville, Ontario
  - Site 1024, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AQX-1125 | Placebo
Started | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — Study Terminated | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AQX-1125 | Placebo | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (6.36) | 50.0 (0.00) | 53.66 (5.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Maximum Daily Pelvic Pain (Mean)
Description: Change from Baseline to Week 12 for AQX-1125 200 mg compared to placebo in the maximum daily pelvic pain score based on a standardized 11-point numeric rating scale (NRS) recorded by electronic diary (eDiary)
Time Frame: 12 Weeks
Population: Study was terminated prematurely, no analysis was performed
Arm/Group | AQX-1125 | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline to Week 12 in NIH-CPSI
Description: Change from Baseline to Week 12 for AQX-1125 200 mg compared to placebo in NIH Chronic Prostatitis Symptom Index (NIH-CPSI) pain subscale and all domains total score
Time Frame: 12 Weeks
Reporting Status: Not Posted

3. Secondary Outcome: Change From Baseline to Week 12 in IIEF-EF
Description: Change from Baseline to Week 12 for AQX-1125 200 mg compared to placebo in Male sexual health as measured using the International Index of Erectile Function Questionnaire, Erectile Function Domain (IIEF-EF)
Time Frame: 12 Weeks
Reporting Status: Not Posted

4. Secondary Outcome: Change From Baseline to Week 12 in Average Daily Pelvic Pain (eDiary),
Description: Change from Baseline to Week 12 for AQX-1125 200 mg compared to placebo in the average daily pelvic pain score based on a standardized 11-point numeric rating scale (NRS) recorded by electronic diary (eDiary)
Time Frame: 12 Weeks
Reporting Status: Not Posted

5. Secondary Outcome: Change From Baseline to Week 12 in Average and Maximum Pelvic Pain Scores in Clinic
Description: Change from Baseline to Week 12 for AQX-1125 200 mg compared to placebo in the average and maximum pelvic pain score based on a standardized 11-point numeric rating scale (NRS) recorded on paper-based questionnaire at clinic visits.
Time Frame: 12 Weeks
Reporting Status: Not Posted

6. Secondary Outcome: Change From Baseline to Week 12 in 24-hour Voiding Frequency (eDiary)
Description: Change from Baseline to Week 12 for AQX-1125 200 mg compared to placebo in voiding frequency as recorded by electronic diary (eDiary)
Time Frame: 12 Weeks
Reporting Status: Not Posted

7. Secondary Outcome: Time Course of Effects From Baseline Through to Week 16: AQX-1125 200 mg Compared to Placebo for Each of the Pain and Symptom Scale Endpoints
Description: Change from Baseline at each clinic visit for AQX-1125 200 mg compared to placebo for; Mean of maximum daily pelvic pain score (eDiary), NIH-CPSI pain subscale and all domains total score, IIEF-EF, Mean of average daily pelvic pain scores (eDiary), average and maximum pelvic pain (Paper-based NRS in clinic), and 24-hour voiding frequency (eDiary)
Time Frame: 16 Weeks
Reporting Status: Not Posted

8. Secondary Outcome: Response to Treatment Compared to Placebo at Week 12 as Measured by the GRA
Description: AQX-1125 200 mg compared to placebo as measured by the Global Response Assessment (GRA) at Week 12
Time Frame: 12 Weeks
Reporting Status: Not Posted

9. Secondary Outcome: Response to Treatment Compared to Placebo at Week 12 as Measured by the PGI-C
Description: AQX-1125 200 mg compared to placebo as measured by the Patient's Global Impression of Change Scale (PGI-C) at Week 12
Time Frame: 12 Weeks
Reporting Status: Not Posted

10. Secondary Outcome: Response to Treatment Compared to Placebo at Week 12 as Measured by the PGI-S
Description: AQX-1125 200 mg compared to placebo as measured by the Patient's Global Impression of Severity Scale (PGI-S) at Week 12
Time Frame: 12 Weeks
Reporting Status: Not Posted

11. Secondary Outcome: The Proportion of Subjects With ≥30% and ≥50% Improvement in Maximum Daily Pelvic Pain Compared to Placebo
Description: Comparison between AQX-1125 200 mg and placebo in proportion of subjects with ≥30% and ≥50% improvement in maximum daily pelvic pain (mean) based on a standardized 11-point numeric rating scale (NRS) recorded by eDiary at Week 6 and 12
Time Frame: 12 Weeks
Reporting Status: Not Posted

12. Secondary Outcome: The Proportion of Subjects With ≥30% and ≥50% Improvement in NIH-CPSI Pain Subscale Compared to Placebo
Description: Comparison between AQX-1125 200 mg and placebo in proportion of subjects with ≥30% and ≥50% improvement NIH-CPSI subscale at Week 6 and 12
Time Frame: 12 Weeks
Reporting Status: Not Posted

13. Secondary Outcome: Response to Treatment
Description: Response to treatment as defined by a decrease in maximum daily pelvic pain (eDiary) at Week 12 with a decrease or no change to concomitant analgesic medication use.
Time Frame: 12 Weeks
Reporting Status: Not Posted

14. Secondary Outcome: Discontinuation of Study Medication Due to Treatment Failure
Time Frame: 12 Weeks
Reporting Status: Not Posted

15. Secondary Outcome: Frequency and Severity of Adverse Events (AEs)
Time Frame: 12 Weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 16 Weeks (12 weeks treatment period and 4 week post last dose follow up)
Arm/Group | AQX-1125 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restrictions are specific to applicable clinical trial agreements with PI(s)

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT03500159/SAP_000.pdf
  • Study Protocol (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/59/NCT03500159/Prot_001.pdf